CLINICAL TRIAL: NCT01383694
Title: Effect of Natural Agonists of TRPV1 in the Treatment of Functional Oropharyngeal Dysphagia in Neurological Diseases and the Elderly: Piperine
Brief Title: Effect Of Piperine In Patients With Oropharyngeal Dysphagia
Acronym: FIS 2009_2
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hospital de Mataró (Other)
Responsible Party: Principal Investigator, Pere Clave, MD, PhD, Hospital de Mataró
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FIS 22/09
Record Dates: First submitted 2011-06-27; First posted 2011-06-28 (Estimated); Last update posted 2015-03-03 (Estimated); Status verified 2015-02

CONDITIONS: Deglutition Disorders
MeSH Terms: conditions — Deglutition Disorders | interventions — piperine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- Piperine Dose 1 (Experimental): Piperine 1 mM
  Interventions: Drug: Piperine
- Piperine Dose 2 (Experimental): Piperine 150 microM
  Interventions: Drug: Piperine

INTERVENTIONS:
Drug: Piperine

SUMMARY:
Piperine acts on the oropharyngeal TRPV1, increasing sensory input and the release of substance P. These actions may accelerate the oropharyngeal swallow response, improving the swallowing of dysphagic patients.

ELIGIBILITY:
Inclusion Criteria:

* Age>18
* History of swallowing difficulties associated with aging and/or neurological diseases (neurodegenerative or non-progressive neurological diseases)
* Study explained and written subject information given
* Informed consent signed

Exclusion Criteria:

* Patients suffering idiosyncratic phenomena or who are allergic to any medication, especially iodinated contrast media
* Patients suffering major respiratory disease or undergoing any type of surgery in the three months prior to the study
* Patients with a background of alcohol dependence or other drug dependence
* Currently participating or having participated in another clinical trial during the last 4 weeks prior to the beginning of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-06; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Safety of swallow | 15 minutes
  Prevalence of penetrations at the laryngeal vestibule

SECONDARY OUTCOMES:
Efficacy of swallow | 15 minutes
  Prevalence of oral and pharyngeal residue

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de Mataró, Mataró, Barcelona, Spain

REFERENCES:
- See also: Publication — http://link.springer.com/article/10.1007%2Fs00535-013-0920-0